CLINICAL TRIAL: NCT03456323
Title: Post-ICU Palliative Care Consultation Intervention Pilot Trial in Older Survivors of Acute Respiratory Failure
Brief Title: Post-ICU Palliative Care Intervention (PIPCI) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAR3202; K23AG045560 (NIH)
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Critical Illness; Frailty; Palliative Care
Keywords: Critical Illness; Frailty; Palliative Care
MeSH Terms: conditions — Critical Illness; Frailty

STUDY DESIGN:
Intervention Model Description: Older survivors of acute respiratory failure and their surrogates (i.e., patient-surrogate pairs, n = 80 participants total) will be randomized to an inpatient palliative care consultation versus usual care in a 1:1 ratio (i.e. 20 patient-surrogate pairs (40 participants total) in each study arm) once enrolled patients are registered to be transferred from the ICU to the general ward.
Who Masked: Outcomes Assessor
Masking Description: The research coordinator who makes the baseline assessment and outcome assessments will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palliative Care Consultation (Experimental): After enrollment the palliative care consultation team will meet with the patient-surrogate pair one or more times to (1) assess symptoms, (2) provide supportive counseling, (3) make symptom treatment recommendations to the primary team of physicians, and (4) will address goals of care.
  Interventions: Behavioral: Palliative Care Consultation
- Usual Care (Placebo Comparator): Patient-surrogate pairs randomized to usual care will continue to receive care by their primary physicians without having a palliative care consultation intervention offered.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Palliative Care Consultation — The palliative care consultation team will be led by one of the board-certified palliative care physicians at Columbia University Medical Center. Over one or more visits, the palliative care consultation team will first review intervention participants' medical records and baseline Edmonton Symptom Assessment System (ESAS) scores. They will also directly assess participants' physical and psychological symptoms. They will provide supportive counseling, make treatment recommendations for burdensome symptoms to the primary team of physicians, and will address goals of care. They will document these activities in structured electronic medical record consultation notes.
  Other Names: PIPCI
  Arms: Palliative Care Consultation
Other: Usual Care — Patient-surrogate pairs randomized to usual care will not have a palliative care consultation intervention offered, and will receive care by their primary physicians. However, if a palliative care consultation is requested after randomization to usual care by the primary team of physicians and/or the patient/surrogate, it will be provided.
  Arms: Usual Care

SUMMARY:
This is a single center, pilot, randomized, single-blind, usual care controlled, pragmatic clinical trial of a post-ICU palliative care consultation intervention in older (age ≥50 years) survivors of acute respiratory failure.

Aim 1: To conduct a pilot post-ICU palliative care consultation intervention trial among frail older ICU survivors and their surrogates. Hypothesis:The Investigators can achieve an adequate enrollment rate, protocol adherence, and intervention fidelity.

Aim 2: To estimate effect sizes and variability for changes in symptoms at hospital discharge and 1 month, and to estimate hospice referral rates and acute-care readmission rates at 1 and 3 months. Hypothesis: Effect sizes and feasibility data will inform and support future post-ICU palliative care studies focused on improving ICU survivorship.

Exploratory Aim. To assess the use of methylphenidate that is recommended and dosed by the palliative care physician for the treatment of moderate-to-severe fatigue. Hypothesis: (1) Not all patients with moderate-to-severe fatigue will be recommended for methylphenidate therapy. (2) Patients prescribed methylphenidate for treatment of moderate-to-severe fatigue after critical illness will adhere to methylphenidate therapy.

DETAILED DESCRIPTION:
There is an urgent need for research to improve outcomes for the rapidly growing population of older survivors of critical illness. Most adults, including older adults, survive critical illness. While recovery with minimal sequelae occurs, a substantial proportion of survivors are left with physical disability and cognitive impairment, have an increased risk of death, and incur high health care costs after hospital discharge. In prior work the Investigators have shown that about 75% of older survivors of respiratory failure are phenotypically frail and that these frail ICU survivors have a high burden of uncontrolled symptoms at hospital discharge and 1-month later. Moderate to severe post-ICU fatigue is the most prevalent symptom and may interfere with functional recovery.

This study is designed to determine whether consultation with a palliative care team may help alleviate any physical symptoms or psychological distress that the patients and their caregivers (surrogates) have coming out of the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years.
* Acute respiratory failure requiring invasive mechanical ventilation, non-invasive mechanical ventilation (continuous or bi-level positive pressure), or high flow nasal cannula for greater than 24 hours in a Columbia University Medical Center medical or surgical ICU.

Exclusion Criteria:

* Hospital discharge directly from ICU.
* Already received palliative care consultation during the hospitalization.
* Planned discharge to hospice or home hospice. These patients do not need further palliative care consultation since they have already decided on prioritizing palliative care over life-sustaining treatment.
* Respiratory failure due to neurologic diagnosis (intracranial hemorrhage, stroke, or coma). These patients are unlikely to be able to participate in any frailty measurements, and may have difficulty with communicating their symptom burden.
* Pre-existing neurologic disease or stroke with motor deficits. Older adults with motor diseases (e.g Parkinson's disease) will be excluded from frailty measurements because they could present with frailty characteristics from a single disease. This criterion was used to exclude subjects in the original Cardiovascular Health Study from which the Fried frailty phenotype was first assessed.
* Psychiatric history of Bipolar Disorder, Schizoaffective Disorder, or Schizophrenia.
* Current Alcoholism or drug abuse.
* Not English or Spanish speaking. Many surveys are not validated in other languages besides English or Spanish. Obtaining interpreters in other languages for palliative care assessments and intervention can be challenging. We expect < 3% of all potentially eligible patients/surrogates to not have English or Spanish speaking ability.
* No healthcare proxy or surrogate also consenting to participate.
* Expected to be discharged to a location >20 miles from Columbia University Medical Center. This discharge radius will make in-person 1-month follow-up feasible.
* Status post heart, lung, or liver transplantation. These patients are not representative of the larger population of older adult survivors of acute respiratory failure.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Annual enrollment rate | 1 year
  The number of patients who enroll compared to the number of patients who enroll and decline enrolling over 1 year
Adherence to the palliative care consultation intervention | From date of Randomization until the date of hospital discharge or 28 days later.
  Proportion of patient-surrogate pairs randomized to a palliative care consultation who actually agree to have the palliative care consultation prior to hospital discharge.
Crossover from usual care to post-ICU palliative care | From date of Randomization until the date of hospital discharge or 28 days later.
  Proportion of patient-surrogate pairs randomized to usual care who end up receiving a post-ICU palliative care consultation prior to hospital discharge.
Fidelity of the palliative care intervention | From date of Randomization until the date of hospital discharge or 28 days later.
  Documentation in electronic medical record consultation notes of (a) burdensome symptoms, (b) supportive counseling, (c) symptom treatment recommendations, and (d) addressing goals-of-care.

SECONDARY OUTCOMES:
Change in Edmonton Symptom Assessment System (ESAS) scores | Pre-randomization baseline until the date of hospital discharge or 28 days later, and 1-month follow-up after hospital discharge.
  Changes in patients' ESAS symptoms (best(0) to worse(10)) from randomization to hospital discharge, and from hospital discharge to 1-month follow-up. ESAS symptoms are: pain, fatigue, drowsiness, nausea, lack of appetite, depression, anxiety, shortness of breath, and wellbeing.
Change in Hospital Anxiety and Depression Scores (HADS) for surrogates | Pre-randomization baseline until the date of hospital discharge or 28 days later, and 1-month follow-up after hospital discharge.
  Changes in surrogates' HADS scores (best(0) to worst(42)) from randomization to hospital discharge, and from hospital discharge to 1-month follow-up.

OTHER OUTCOMES:
Number of patients with moderate-to-severe fatigue who are recommended for and receive methylphenidate treatment. | Randomization until 1-month follow-up after hospital discharge.
  Number of patients with ESAS fatigue scores greater than or equal to 4 at baseline who are recommended for and receive methylphenidate treatment.
New limitation of life-sustaining therapy | Day of hospital discharge until 3-month follow-up after hospital discharge.
  Number of patients who elect DNR after randomization
Enrollment in Hospice | Day of hospital discharge until 3-month follow-up after hospital discharge.
  Number of patients who enroll in-patient hospice or home hospice.
Acute-care readmissions | Day of hospital discharge until 3-month follow-up after hospital discharge.
  Number of patients who are re-admitted to an acute care hospital within 1-month and 3-months.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Baldwin, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No